CLINICAL TRIAL: NCT01397071
Title: Hass Avocado Flesh Inhibition of Appearance of Lipid Peroxidation Products When Added to a Ground Beef Patty Consumed by Healthy Volunteers
Brief Title: Effects of Avocado When Added to a Meat Patty on Inflammation in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HAB-001
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
Keywords: Avocado, antioxidant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ground Beef Patty with Avocado (Active Comparator): Test burgers with fresh avocado added just prior to consumption
  Interventions: Other: Avocado
- Ground Beef Patty without Avocado (Active Comparator): Test burgers
  Interventions: Other: Avocado

INTERVENTIONS:
Other: Avocado — Fresh Avocado

SUMMARY:
Avocados are naturally rich in antioxidants, or beneficial compounds, that can help prevent many diseases, like atherosclerosis (hardening of the arteries). When foods that are high in fats are eaten, certain harmful compounds can be absorbed, which can lead to atherosclerosis. One harmful compound is called malondialdehyde, or MDA. This compound can be measured in the blood and the urine after a person eats a high fat meal. Antioxidants found in herbs and spices may lower the absorption of MDA, which could help prevent the development of atherosclerosis.

This study will determine whether the beneficial compounds of avocado can reduce absorption of MDA. This will be tested by asking healthy males to eat a high fat ground beef patty with or without avocado and then measuring the amount of MDA in their blood and urine samples. Blood flow will also be measured. Healthy men have been chosen for this study because eating high fat hamburger patties can easily mimic in them the condition that causes atherosclerosis. Avocados are rich in antioxidants, which have been shown in previous studies to reduce the absorption of harmful compounds, like MDA, that are formed during cooking. The results from this study may help to explain how high fat foods can be harmful to the body and how beneficial antioxidants from herbs and spices can protect the body.

This will be determined from blood and urine samples after the subjects are given two different meals: a) a plain cooked ground beef patty, and b) or avocado with a cooked ground beef patty.

DETAILED DESCRIPTION:
The Hass Avocado contains monounsaturated fat, lutein, glutathione, vitamin E, and other antioxidants. This study will determine whether avocado exerts a beneficial effect by inhibition of the absorption of malondialdehyde (MDA) which is a measure of lipid peroxidation. In a previous study, we demonstrated that spice antioxidants resulted in a 70 percent decrease in the formation of MDA during cooking and that healthy volunteers consuming burgers made with spice excreted 50 percent less MDA in their urine than subjects consuming a control burger made without spices. Since the spices were added during cooking of the burger, it was not possible to assess the effects of the antioxidants in the stomach. Foods in the stomach continue to form lipid peroxidation products during digestion and this is called the "bioreactor" function of the stomach. In the proposed study known quantities of fresh avocado will be placed on top of a burger prior to consumption to determine whether the avocado inhibits formation of MDA from cooked burger meat in the stomach. Study demonstrated an increase in inflammatory and oxidative markers in mononuclear cells using Western blot analysis of nuclear factor-kappa light chain enhancer of activated B cells (NFkB) and NADPH oxidase subunits following a mixed high calorie meal. Considering the rich content of bioactive compounds in the avocado, we therefore selected these methods for the endpoint determinations as well in this proposed randomized, crossover study.

We will accomplish the following specific aims:

1. To measure plasma and urine malondialdehyde by high performance liquid chromatography before and over6 hours after consumption of the test burgers with or without fresh avocado added just prior to consumption.
2. To measure insulin, glucose, triglycerides, tumor necrosis factor alpha (TNF-α), interleukin 6 (IL-6), Interleukin 8 (IL-8), NFkB activation, nitric oxide and peripheral arterial tonometry after each test burger.

These studies will add to the evidence that antioxidants in a lipid phase can inhibit formation and/or absorption of cytotoxic lipid products such as malondialdehyde. Ultimately, a better understanding of the role of bioactive substances from plant foods such as the avocado may demonstrate the importance of plant-based antioxidants in human health.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 35 years old males (inclusive)
* Non-smokers
* Must weigh a minimum of 110 pounds
* Willing to maintain normal activity and eating patterns for the duration of the study
* Willing to maintain their normal diet for the duration of the study but avoid dairy, avocado and meat products.

Exclusion Criteria:

* Females
* Abnormal liver function (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2 x upper limit)
* Currently taking steroidal drugs
* Known HIV positive or AIDS
* Chronic infectious disease
* Cancer treated within the past two years
* Participation in a therapeutic research study within 30 days of baseline
* Consumption of vegetarian diet
* Allergy or sensitivity to dairy products
* Allergic to avocado

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Heber, MD, PhD, Principal Investigator — UCLA Center for Human Nutrition
Locations (1):
- UCLA Center for Human Nutriiton, Los Angeles, California, United States

REFERENCES:
- [Result] Li Z, Wong A, Henning SM, Zhang Y, Jones A, Zerlin A, Thames G, Bowerman S, Tseng CH, Heber D. Hass avocado modulates postprandial vascular reactivity and postprandial inflammatory responses to a hamburger meal in healthy volunteers. Food Funct. 2013 Feb 26;4(3):384-91. doi: 10.1039/c2fo30226h. PMID 23196671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period was 8/2011 to 2/2012. Enrollment took place in a private setting in the clinic located at the site.
Pre-assignment Details: 17 healthy male volunteers were recruited and screened; 6 failed screen; 11 participants completed crossover study.
Groups:
- Consumption of Beef Patty With or Without Avocado Added: Participants consumed 250 g cooked ground beef patty with or without avocado added prior to ingestion.
Period: Consumption of Beef Patty Alone
Arm/Group | Consumption of Beef Patty With or Without Avocado Added
Started | 11
Completed | 11
Not Completed | 0
Period: Consumption of Beef Patty With Avocado
Arm/Group | Consumption of Beef Patty With or Without Avocado Added
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Consumption of Beef Patty With or Without Avocado: Participants consumed 250 g cooked ground beef patty with or without 68 g fresh avocado added prior to ingestion.
Arm/Group | Consumption of Beef Patty With or Without Avocado
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (5.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male participants | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black | 2
  White | 4
  Hispanic | 4
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change of Endothelial Function by Measurement of Flow-mediated Vasodilation Using the Reactive Hyperemia Index (RHI)
Description: Change from baseline in reactive hyperemia index (RHI) in response to consumption of 250 g beef patty with or without 68 g avocado added at 2 hour post-ingestion. RHI is a measure of endothelial dysfunction using noninvasive peripheral arterial tonometry (PAT). It is a ratio of the post-to-pre occlusion PAT amplitude of the tested arm, divided by the post-to-pre occlusion ratio of the control arm. RHI less than 1.67 is considered sign of endothelial dysfunction and RHI equal to or greater than 1.67 is considered normal function. The possible range of scores is 1 to 3. Increasing score indicates the improvement of coronary endothelial function.
Time Frame: Baseline and 2 hours post-ingestion
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Participants Consumed 250 g Beef Patties Alone: Participants consumed 250 g beef patties without avocado added
- Participants Consumed 250 g Beef Patties With Avocado Added: Participants consumed 250 g beef patties with 68 g avocado added prior to ingestion.
Arm/Group | Participants Consumed 250 g Beef Patties Alone | Participants Consumed 250 g Beef Patties With Avocado Added
Number analyzed (Participants) | 11 | 11
score on a scale
  PAT index before intervention | 2.20 (0.36) | 2.17 (0.57)
  PAT index at 2 hr after intervention | 1.56 (0.21) | 2.08 (0.51)
Statistical Analysis 1: Comparison: Participants Consumed 250 g Beef Patties Alone vs Participants Consumed 250 g Beef Patties With Avocado Added; Comparison of change in PAT measurements was made to beef alone vs. beef with avocado 2 hours post-ingestion; Test type: Other; p = 0.052, t-test, 2 sided; Mean Difference (Final Values) = 2.20

2. Secondary Outcome: Change in Inflammation Marker Nuclear Factor of Kappa Light Polypeptide Gene Enhancer in B-cells Inhibitor Alpha (IkB-alpha)
Description: Change from baseline inflammatory marker IkB-alpha in response to the consumption of 250 g beef patty with or without 68 g avocado added was assessed at 0 (baseline), 1, 2, 3, 4, 5, 6 hours post-ingestion. Baseline and 3 hours post-ingestion was reported.
Time Frame: 0 (baseline) and 3 hours post-ingestion
Measure: Mean (Standard Deviation); unit: percentage of baseline
Groups:
- Consumption of Beef Patty Alone: Participants consumed 250 g beef patties without avocado added prior to ingestion.
- Consumption of 250 g Beef Patty With Avocado Added: Participants consumed 250 g beef patties with 68 g avocado added prior to ingestion.
Arm/Group | Consumption of Beef Patty Alone | Consumption of 250 g Beef Patty With Avocado Added
Number analyzed (Participants) | 11 | 11
percentage of baseline
  IkB-alpha at baseline | 100 (0.0) | 100 (0.0)
  IkB-alpha 3 h after intervention | 57.8 (15) | 131.3 (26.8)
Statistical Analysis 1: Comparison: Consumption of Beef Patty Alone vs Consumption of 250 g Beef Patty With Avocado Added; Comparison was made to beef patty alone vs. beef patty with avocado added 3 hours post-ingestion; Test type: Other; p = 0.03, t-test, 2 sided — Significance is defined as p<0.05; % of baseline = 0.58

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 3 months period
Description: Participants were monitored and questioned regarding the occurrence and nature of any adverse experiences.
Groups:
- Change in PAT After Consuming Beef Only: Change in peripheral arterial tonometry (PAT) after consuming meals consisting of a ground beef patty only.
- Change in PAT After Comsuming Beef With Avocado: Change in peripheral arterial tonometry (PAT) after consuming meals consisting of a ground beef patty with 68 grams of avocado added.
Arm/Group | Change in PAT After Consuming Beef Only | Change in PAT After Comsuming Beef With Avocado
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No